CLINICAL TRIAL: NCT03362385
Title: Impact of Obstructive Sleep Apnea and Continuous Positive Airway Pressure Therapy on Outcomes in Patients With Acute Coronary Syndrome: The OSA-ACS Project
Brief Title: OSA-ACS Project: Association of OSA and CPAP Therapy With Outcomes in ACS Patients
Status: Completed | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Shao-Ping Nie, Director, Emergency & Critical Care Center, Professor of Medicine, Beijing Anzhen Hospital
Other Study IDs: 2013025
Record Dates: First submitted 2017-11-07; First posted 2017-12-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Obstructive Sleep Apnea of Adult; Acute Coronary Syndrome
Keywords: Obstructive sleep apnea; Acute coronary syndrome; Continuous positive airway pressure; Outcome
MeSH Terms: conditions — Acute Coronary Syndrome; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OSA
  Interventions: Other: Patients with OSA based on sleep study
- Non-OSA
  Interventions: Other: Patients without OSA based on sleep study

INTERVENTIONS:
Other: Patients with OSA based on sleep study — Polysomnography or Polygraphy
  Groups: OSA
Other: Patients without OSA based on sleep study — Polysomnography or Polygraphy
  Groups: Non-OSA

SUMMARY:
Obstructive sleep apnea (OSA) is an increasingly common chronic disorder in adults that has been strongly associated with various forms of cardiovascular disease. Compared to the general population, OSA occurs more often in patients with acute coronary syndrome (ACS). Although percutaneous coronary intervention (PCI) is nowadays part of standard therapy and optimal medical therapy has been used to manage traditional risk factors, the long-term cardiovascular outcomes after index ACS remain suboptimal.

Some preliminary data suggest OSA is associated with higher risk of subsequent cardiovascular events in ACS patients. However, the study population was heterogeneous and these studies were not done in the context of new-generation drug-eluting stents and intensive antiplatelet therapy, thus precluding definite conclusions. Furthermore, a cardioprotective role of OSA in the context of acute myocardial infarction (AMI), via ischemic preconditioning, has also been postulated.

Due to the inconsistent evidence, the investigators performed a large-scale, prospective cohort study to delineate the whole picture of the association of OSA with short- and long-term outcomes of patients with ACS. Whether treatment of OSA (eg. continuous positive airway pressure (CPAP)) would prevent these events will also be evaluated. Moreover, the investigators will assess the potential mechanisms of OSA-induced atherosclerosis and myocardial injury in ACS patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Admission with an ACS (including STEMI, NSTEMI, and unstable angina)
3. Written informed consent

Exclusion Criteria:

1. Cardiogenic shock (systolic blood pressure <90mmHg)
2. Cardiac arrest on admission or during hospitalization
3. Severe insomnia, chronic sleep deprivation, abnormal circadian rhythm (sleep duration <4h/night)
4. Predominantly central sleep apnea (CSA, ≥50% central events or central apnea hypopnea index (AHI) ≥10/h)
5. Previous or current use of CPAP
6. Known or planned pregnancy
7. Severe comorbidities: eg. malignancy (life expectancy <2 years)
8. Patients who cannot tolerate the sleep study or refuse it

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In-hospital patients with ACS and undergoing sleep study
Sampling Method: Non-Probability Sample
Enrollment: 2160 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac and cerebrovascular events (MACCEs) | Median 24 months
  Including cardiovascular death, myocardial infarction, stroke, ischemia-driven revascularization, and hospitalization for unstable angina or heart failure

SECONDARY OUTCOMES:
Cardiovascular death | Median 24 months
All-cause mortality | Median 24 months
Hospitalization for unstable angina | Median 24 months
Ischemia-driven revascularization | Median 24 months
Any repeat revascularization | Median 24 months
Myocardial salvage index (assessed by CMR) | 3 months
Relative proliferation volume within stent segment (% of stent volume) | 12 months
MACCEs | Median 24 months
  Effect of continuous positive airway pressure (CPAP) treatment on MACCEs in patients with OSA and ACS

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, China

REFERENCES:
- [Derived] Qiu Y, Li Z, Hao W, Liu X, Guo Q, Guo Y, Que B, Gong W, Zheng W, Wang X, Nie S. Association of Obstructive Sleep Apnea With Cardiovascular Events in Acute Coronary Syndrome Patients With or Without Excessive Daytime Sleepiness: A Prospective Cohort Study. Rev Cardiovasc Med. 2025 Jul 28;26(7):33439. doi: 10.31083/RCM33439. eCollection 2025 Jul. PMID 40776960
- [Derived] Zhang Y, Xu D, Zheng W, Hao W, Zhen L, Yan Y, Wang X, Nie S. Impact of Obstructive Sleep Apnea and Triglyceride Glucose Index on Cardiovascular Events in Acute Coronary Syndrome Patients: A Post-Hoc Analysis of the OSA-ACS Study. Rev Cardiovasc Med. 2025 May 21;26(5):36205. doi: 10.31083/RCM36205. eCollection 2025 May. PMID 40475723
- [Derived] Zhou Y, Gong W, Yan Y, Wang X, Zheng W, Que B, Li S, Zhang Z, Chen X, Fan J, Zhao W, Xin Q, Ai H, Nie S. Prognostic implications of obstructive sleep apnea in patients with unstable angina stratified by remnant cholesterol and triglyceride: a prospective cohort study. BMC Cardiovasc Disord. 2024 Oct 12;24(1):549. doi: 10.1186/s12872-024-04214-1. PMID 39395961
- [Derived] Zhang Z, Ai H, Yan M, Zheng W, Yan Y, Wang X, Fan J, Que B, Li S, Wang G, Gong W, Nie S. Prognostic effect of obstructive sleep apnea in acute coronary syndrome patients with heart failure. Respir Med. 2024 Nov-Dec;234:107814. doi: 10.1016/j.rmed.2024.107814. Epub 2024 Sep 21. PMID 39307479
- [Derived] Chen X, Zhen L, Ai H, Que B, Fan J, Wang X, Yan Y, Li S, Zhang Z, Zhou Y, Gong W, Nie S. Prognostic implications of obstructive sleep apnea in patients with acute coronary syndrome stratified by homocysteine level: a prospective cohort study. Respir Res. 2023 Dec 14;24(1):313. doi: 10.1186/s12931-023-02627-8. PMID 38098080
- [Derived] Wang G, Miao H, Hao W, Zhao G, Yan Y, Gong W, Fan J, Ai H, Que B, Wang X, Nie S. Association of obstructive sleep apnoea with long-term cardiovascular events in patients with acute coronary syndrome with or without hypertension: insight from the OSA-ACS project. BMJ Open Respir Res. 2023 Jun;10(1):e001662. doi: 10.1136/bmjresp-2023-001662. PMID 37369551
- [Derived] Wang B, Hao W, Fan J, Yan Y, Gong W, Zheng W, Que B, Ai H, Wang X, Nie S. Clinical significance of obstructive sleep apnea in patients with acute coronary syndrome with or without prior stroke: a prospective cohort study. Eur J Med Res. 2023 Mar 1;28(1):107. doi: 10.1186/s40001-023-01071-0. PMID 36859391
- [Derived] Hao W, Wang X, Fan J, Guo R, Gong W, Yan Y, Zheng W, Que B, Ai H, Ma C, Ma X, Nie S. Prognostic Implications of OSA in Acute Coronary Syndrome by Obesity Status. Chest. 2023 Jul;164(1):219-230. doi: 10.1016/j.chest.2023.02.001. Epub 2023 Feb 9. PMID 36764513
- [Derived] Li Z, Miao H, Zhang S, Fan J, Yan Y, Gong W, Zheng W, Wang X, Que B, Ai H, Zhang L, Nie S. The value of nurse-led anthropometric and oropharyngeal measurements combined with STOP-Bang questionnaire in screening for obstructive sleep apnea in patients with acute coronary syndrome: a prospective cohort study. BMC Pulm Med. 2022 Nov 3;22(1):396. doi: 10.1186/s12890-022-02200-x. PMID 36329414
- [Derived] Lv Q, Jiao X, Yu H, Sun Q, Li F, Wang Y, Sun H, Du Z, Li L, Hu C, Zhang M, Nie S, Qin Y. ANGPTL3 and Cardiovascular Outcomes in Patients With Acute Coronary Syndrome and Obstructive Sleep Apnea. J Am Heart Assoc. 2022 Sep 20;11(18):e025955. doi: 10.1161/JAHA.122.025955. Epub 2022 Sep 8. PMID 36073641
- [Derived] Zeng Y, Yang S, Wang X, Fan J, Nie S, Wei Y. Prognostic impact of residual SYNTAX score in patients with obstructive sleep apnea and acute coronary syndrome: a prospective cohort study. Respir Res. 2019 Feb 28;20(1):43. doi: 10.1186/s12931-019-1008-z. PMID 30819182
- [Derived] Zhou SH, Wang X, Fan JY, Gong W, Zhao GQ, Hao W, Li AB, Guo RF, Shi H, Li ZX, Nie SP, Wei YX. [Prospective cohort study on the impact of moderate/severe obstructive sleep apnea on the prognosis of patients with acute myocardial infarction]. Zhonghua Xin Xue Guan Bing Za Zhi. 2018 Aug 24;46(8):622-628. doi: 10.3760/cma.j.issn.0253-3758.2018.08.009. Chinese. PMID 30139013
- [Derived] Zhao GQ, Wang X, Fan JY, Gong W, Hao W, Zhou SH, Li AB, Guo RF, Shi H, Li ZX, Nie SP, Wei YX. [Association between hypothyroidism and sleep breathing disorders in patients with coronary heart disease]. Zhonghua Nei Ke Za Zhi. 2018 Aug 1;57(8):571-575. doi: 10.3760/cma.j.issn.0578-1426.2018.08.007. Chinese. PMID 30060328